CLINICAL TRIAL: NCT06766643
Title: A Prospective, Randomized, Controlled Phase II Clinical Trial of Stereotactic Radiosurgery Versus Radiofrequency Ablation in Primary Liver Cancer in a Special Site of Surgical Evaluation for Non-operable
Brief Title: Stereotactic Radiosurgery Versus Radiofrequency Ablation for Primary Liver Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241490
Record Dates: First submitted 2024-12-22; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Primary Liver Cancer
Keywords: Primary liver cancer，Stereotactic body radiation therapy，Radiofrequency ablation therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic body radiation therapy group (Experimental)
  Interventions: Procedure: Stereotactic Body Radiation Therapy (SBRT)
- Radiofrequency ablation therapy group (Experimental)
  Interventions: Procedure: Radiofrequency ablation therapy

INTERVENTIONS:
Procedure: Stereotactic Body Radiation Therapy (SBRT) — Stereotactic radiosurgery for liver lesions: with a total dose of 40~50Gy/3~5fraction;
  Arms: Stereotactic body radiation therapy group
Procedure: Radiofrequency ablation therapy — Radiofrequency ablation therapy:1 complete radiofrequency ablation of liver lesions for liver lesions
  Arms: Radiofrequency ablation therapy group

SUMMARY:
A phase II clinical trial of stereotactic radiosurgery versus radiofrequency ablation in the treatment of inoperable primary liver cancer in specific sites

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled Phase II clinical trial aimed at recruiting patients with primary liver cancer who are deemed inoperable after surgical evaluation, with tumor lesions located near major blood vessels, the diaphragm, the liver capsule, or the porta hepatis. The objective of this study is to evaluate the efficacy and safety of stereotactic radiotherapy and radiofrequency ablation as treatment options for such patients. It must be determined by the investigator whether stereotactic radiotherapy or radiofrequency ablation is the preferred treatment for these patients. Eligible patients will be randomly assigned in a 1:1 ratio to one of the following treatment groups: stereotactic radiotherapy or radiofrequency ablation. The study is expected to enroll 65 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to implementing any trial-related procedures, written informed consent must be signed;
2. Age ≥ 18 years and ≤ 75 years;
3. Child-Pugh score ≤ 7;KPS score ≥ 70;
4. The patient must be clearly diagnosed with hepatocellular carcinoma, usually confirmed through imaging (CT, MRI) or histological examination (biopsy);
5. The tumor is located near major blood vessels/diaphragm/liver capsule/liver hilum;
6. Surgically assessed as inoperable hepatocellular carcinoma or recurrence of primary hepatocellular carcinoma within 2 years after radical treatment;
7. According to the criteria for evaluating the efficacy of solid tumors, there should be at least one measurable lesion by imaging, with the lesion size not exceeding 5 cm; total number of lesions ≤ 3;
8. No previous anti-tumor treatment;
9. Normal liver (liver volume minus tumor volume) is sufficient;
10. Normal major organ functions, including blood routine tests [absolute neutrophil count (ANC) ≥ 1.5 × 10^9, platelets ≥ 70 × 10^9, hemoglobin ≥ 80 g/L], liver function tests [bilirubin < 3.0 mg/dL, international normalized ratio (INR) < 1.7, albumin ≥ 2.8 g/dL, aspartate transaminase (AST)/alanine transaminase (ALT) < 6], serum creatinine < 1.5 times the upper limit of normal, or creatinine clearance ≥ 60 mL/min;
11. Stable respiration for more than 10 minutes;
12. Expected survival time > 2 years.

Exclusion Criteria:

1. Possible surgical intervention;
2. Presence of other serious comorbidities, such as uncontrolled cardiovascular diseases, pulmonary diseases, or dysfunction of other organs, where the overall health status is poor and may result in treatment intolerance;
3. Severe liver dysfunction exceeding the specific criteria defined in the trial;
4. Other malignancies diagnosed within 5 years prior to the first treatment or at the time of diagnosis of hepatocellular carcinoma;
5. Significant clinically meaningful bleeding symptoms or a clear bleeding tendency within 3 months prior to enrollment;
6. Currently participating in an interventional clinical trial treatment, or having received other investigational drugs or used investigational devices within 4 weeks before the first treatment;
7. Previous treatment with anti-target tumor therapies;
8. History of upper abdominal radiotherapy;
9. Uncontrolled active comorbidities;
10. Not meeting the expected survival prognosis or unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Until the end of the study, about 2 years

SECONDARY OUTCOMES:
Overall survival rate | Until the end of the study, about 2 years
Local control rate | Until the end of the study, about 2 years
Intrahepatic control rate | Until the end of the study, about 2 years
Extrahepatic control rate | Until the end of the study, about 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobiliary Oncology and Radiation Oncology,Tianjin Medical University Cancer Institute & Hospital,Key Laboratory of Cancer Prevention and Therapy,National Clinical Research Center for Cancer, Tianjin's Clinical Research Center for Cancer, Tianjin, China